CLINICAL TRIAL: NCT04976153
Title: Skeletal Muscle-derived Cell Implantation for the Treatment of Fecal Incontinence: a Phase III, Randomized, Controlled, Double Blind, Two Armed Clinical Study
Brief Title: Skeletal Muscle-derived Cell Implantation for Treatment of Fecal Incontinence
Acronym: Fidelia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Innovacell GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IC-01-02-5-009
Record Dates: First submitted 2021-07-05; First posted 2021-07-26 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- aSMDC (Experimental): Autologous skeletal muscle derived cells for the treatment of urge fecal incontinence
  Interventions: Biological: aSMDC
- Placebo (Placebo Comparator): Placebo control is the vehicle solution used for the study product
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: aSMDC — Autologous Muscle Derived Cells for injection into the external anal sphincter
  Arms: aSMDC
Other: Placebo — Placebo control is the vehicle solution used for the study product
  Arms: Placebo

SUMMARY:
The objective of this study is the final assessment of clinical safety and efficacy of autologous autologous skeletal muscle derived cells for patients with urge fecal incontinence due to external anal sphincter dysfunction caused by its disruption and/or weakness.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years old
* Patients who are mentally competent and able to understand all study requirements
* Female patients of childbearing potential willing to use appropriate methods of contraception
* Patient has symptoms of urge fecal incontinence with a disease duration of at least 6 months and did not improve sufficiently by conservative treatment performed for at least 3 months
* Urge fecal incontinence episodes that occur more than twice a week
* Maximal incremental voluntary squeeze pressure (increase to resting pressure) on anal manometry is 100mmHg or less in women and 150mmHg or less in men
* 9. Ultrasound of the anal canal showing intact external anal sphincter or a maximal overall extent of external anal sphincter injury and tear of 180 degrees

Exclusion Criteria:

* Patients for whom the investigator determines that FI has a different cause than external anal sphincter dysfunction.
* Patients with global fragmentation of the external anal sphincter as assessed by anal canal ultrasound
* Patients who underwent any anorectal surgery within 6 months before screening visit
* Patients who underwent a total of two or more external anal sphincter-related surgeries
* Patients who currently have anal fistulas or fissures or have recurrent anal fistulas or fissures
* Patients with poorly controlled chronic constipation including obstructed defecation syndrome
* Patients with indications against a surgery under anesthesia
* Patients with a malignant disease not in remission for 5 years or more
* Patients who have undergone radiation therapy of the bowel and pelvis
* Patients who have undergone chemotherapy within last 5 years prior to study enrolment and/or chemotherapy related neuropathy of the bowel and pelvis
* Patients with compromised immune system and/or rheumatic disease, and patients under immunosuppressive therapy
* Patients with a diagnosis of chronic inflammatory bowel disease (e.g Crohn's disease, Colitis Ulcerosa)
* Patients suffering from a disease which has not been resolved within 4 weeks prior to screening including fever and/or diarrhea of unknown reasons (4 weeks)
* Patients diagnosed with human immunodeficiency virus (HIV), acute or chronic viral hepatitis HCV, acute or chronic viral hepatitis HBV, active Syphilis or HTLV (tested upon risk assessment by investigator)
* Patients diagnosed with any kind of skeletal muscle disease and/or neuronal disorders
* Patients with severe myocardial disorders, irregular pulse or a pacemaker
* Patients with implantations of metal components in the electrical stimulation treatment area
* Patients with uncontrolled diabetes mellitus type I or II, or suffering from diabetic peripheral neuropathic pain
* Patients with clinically relevant abnormal laboratory values judged by the responsible investigator as relevant for the study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in frequency of incontinence episodes | 12 Months
  Urge fecal incontinence

CONTACTS AND LOCATIONS:
Locations (31):
- Austria (2):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Medical University Graz, Graz
- Medical Center Unimed EOOD, Sevlievo, Bulgaria
- Czechia (2):
  - Fakultni nem. u sv. Anny v Brne, Brno, Brno
  - The Institute for the Care of Mother and Child, Prague
- France (4):
  - Deaconess Hospital Group Croix Saint - Simon, Paris, France
  - Hospital Bichat - Claude Bernard, Paris, France
  - CHU Rennes - Hospital Pontchaillou, Rennes
  - CHU de Rouen, Rouen
- Heidelberg University, Medical Faculty Mannheim, Department of surgery, Mannheim, Germany
- IRCCS Ospedale San Raffaele, San Donato Milanese, Italy
- Japan (11):
  - Hokkaido Railway Company JR Sapporo Hospital, Sapporo, Hokkaido
  - Tsujinaka Hospital, Coloproctological Surgery, Chiba
  - Teikyo University Chiba Medical Center, Chiba
  - Kurume Hospital, Fukuoka
  - Hiroshima Memorial Hospital, Hiroshima
  - Meiwa Hospital, Hyōgo
  - Matsushima Hospital, Kanagawa
  - Coloproctology Center Takano Hospital, Kumamoto
  - Japan Post Kyoto Teishin Hospital, Kyoto
  - Jichi Medical University Hospital, Tochigi
  - Juntendo University Hospital, Tokyo
- Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie, Krakow, Poland
- Spain (4):
  - Corporacio Sanitaria Parc Tauli, Barcelona
  - Hospital de Mataro, Mataró
  - Hosp. General Universitario Morales Meseguer, Murcia
  - Luis Garcia Florez, Oviedo
- Sweden (3):
  - Skånes Universitetssjukhus, Malmo, Malmo, Sweden
  - Östersund sjukhus, Kirurgiska kliniken, Östersund, Sweden
  - Danderyd Sjukhus, Danderyd
- St. Mary's Hospital, London, United Kingdom